CLINICAL TRIAL: NCT06714773
Title: Grade 2 Chondrosarcoma Treated by Intralesional Curettage: Follow-up vs Resection
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: CONDRO2
Record Dates: First submitted 2024-11-28; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-10

CONDITIONS: Chondrosarcoma, Grade 2
Keywords: intralesional curettage
MeSH Terms: conditions — Chondrosarcoma; Lymphoma, Follicular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to assess the oncological outcomes in patients diagnosed with grade 2 chondrosarcoma, treated with intralesional curettage, stratified into two cohorts: those subjected to follow up monitoring and those who have undergone subsequent surgical intervention.

DETAILED DESCRIPTION:
Large resection of the tumor is considered the treatment of choice in patients affected by grade 2 chondrosarcoma. Nonetheless, a preoperative diagnosis of a lower grade lesion (ChS grade 1) is not infrequent, thus making these patients treated with intralesional curettage. Intralesional curettage is a type of surgery in which the pathological component is removed from the affected bone and the resulting bone defects can be filled with bone substitutes or bone cement. Bone cortexes are left in place like a shell.

The results of this study could contribute to find the right therapeutic pathway in patients affected by grade 2 chondrosarcoma treated with intralesional curettage, in particular in patients who underwent further surgery (bone resection) or follow-up. Since outcome data are scarce in the literature, the results of this study could be used to assess the feasibility of a randomized controlled trial with the correct sample size.

It is an explorative, spontaneous, non-profit, retrospective, observational study.

It involves the pseudonymous data collection of all patients matching inclusion criteria. The data recorded in this study are extracted from the medical records of patients who regularly seek care from the medical unit during their routine clinical visits. Following a meticulous collection of patients' baseline data, the two therapeutic options (clinical monitoring or bone resection) in patients affected by grade 2 chondrosarcoma treated with intralesional curettage will be compared.

Data related to demographics, histologic and treatment data will be collected. Oncologic follow-up data will be also collected. In particular, data related to local recurrences, distant metastasis and survival will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of grade 2 chondrosarcoma of the appendiceal skeleton in the definitive specimen;
* Patients treated with intralesional curettage surgery;
* Patients aged >=18 years;
* Patients who were treated between 01/01/2008 and 31/12/2020.

Exclusion Criteria:

* Patients diagnosed with grade 1 or 3 chondrosarcoma on the histological diagnosis of the operative specimen.
* Patients undergoing wide resection as the primary treatment.
* Patients with less than 12 months follow-up.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All adult patients with diagnosis of grade 2 chondrosarcoma of the appendiceal skeleton who underwent intralesional curettage surgery, treated between 01/01/2008 and 31/12/2020.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-01-20 (Actual); Primary Completion 2024-07-20 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Tumor recurrence(%) | 3 months, 6 months, 1 year, 2 years, 5 years, 10 years
  It will be measured by: X-Rays, CT, MRI, PET CT scan
distant metastasis (%) | 3 months, 6 months, 1 year, 2 years, 5 years, 10 years
  It will be measured by: CT scan of the lungs, PET CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Sambri, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Italy